CLINICAL TRIAL: NCT03470909
Title: SKINI - Prospective Evaluation of the Radicality of Breast Tissue Removal With Skin-Sparing and Nipple-Sparing Mastectomy (SSM or NSM)
Brief Title: SKINI - Radicality of Skin-Sparing and Nipple-Sparing Mastectomy
Acronym: SKINI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brust-Zentrum AG (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-01191
Record Dates: First submitted 2018-03-05; First posted 2018-03-20 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Surgery
Keywords: Remaining breast tissue; Skin-Sparing Mastectomy; Nipple-Sparing Mastectomy; Prophylactic
MeSH Terms: interventions — Mastectomy, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin-Sparing Mastectomy (SSM) (Other)
  Interventions: Procedure: Skin-Sparing Mastectomy (SSM)
- Nipple-Sparing Mastectomy (NSM) (Other)
  Interventions: Procedure: Nipple-Sparing Mastectomy (NSM)

INTERVENTIONS:
Procedure: Skin-Sparing Mastectomy (SSM) — For patients undergoing SSM, 10 points of interest in radial localization have been selected for investigation of the presence of residual breast tissue.
  The points are located under the remaining skin envelope and will be investigated by performing small biopsies with a cervical biopsy forceps.
  Additionally, the distance between the surface of the specimen and the glandular tissue will be explored at five points at the base of the removed breast.
  These histological sections will be radially oriented.
  Arms: Skin-Sparing Mastectomy (SSM)
Procedure: Nipple-Sparing Mastectomy (NSM) — For patients undergoing NSM, 14 points of interest in radial localization have been selected for investigation of the presence of residual breast tissue, i.e. comparing to SSM, 4 additional biopsies will be taken behind the peripheral part of the areola.
  The points are located under the remaining skin envelope and will be investigated by performing small biopsies with a cervical biopsy forceps.
  Additionally, the distance between the surface of the specimen and the glandular tissue will be explored at five points at the base of the removed breast.
  These histological sections will be radially oriented.
  Arms: Nipple-Sparing Mastectomy (NSM)

SUMMARY:
Prospective collection of health related personal data and biological material (tissue biopsy) in patients undergoing mastectomy.

DETAILED DESCRIPTION:
In this prospective, multi-center trial patients undergoing mastectomy and fulfilling inclusion criteria receive additional biopsies from the remaining skin envelope in order to quantify the amount of residual breast tissue.

Since the investigators will assess, 142 breasts will be investigated. This means a maximum of n=142 patients will be included (corresponding to a minimum of n=71 patient).

On the specimen additional histological sections in radial direction will be performed.

The aim of the study is to evaluate the quality of Skin- Sparing and Nipple-Sparing Mastectomy. On each predefined location in the wound cavity the investigators will investigate where residual breast tissue (RBT) will be found or not. If no RBT can be detected at all predefined breast locations this breast will be classified as having no RBT (=RBT negative). If breast tissue can be detected the investigators have a RBT positive breast.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing uni- or bilateral Skin-Sparing or Nipple-Sparing mastectomy
* Female participants ≥ 18 years of age
* The subject was informed on the project and gave her written informed consent to use her data and samples for this project.

Exclusion Criteria:

- Not fulfilling inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
Detection of residual breast tissue (RBT) | 20 months
  Each biopsy specimen will be histopathologically assessed for the presence of residual breast tissue (RBT), i.e. in case of SSM 10 biopsy specimens (points A-K) and in case of NSM 14 biopsy specimens (points A-O).
  A mastectomy is defined as RBT-positive whenever residual breast tissue will be detected in one or more biopsies. RBT will be assessed as binary dependent variable (0: no RBT; 1: at least one probe with positive breast tissue detection) and correlated with patient- and therapy-related factors, including age, BMI, breast weight, side of mastectomy (left vs. right), type of mastectomy (SSM vs. NSM), skin flap necrosis, indication for mastectomy, axilla surgery, preoperative treatment, surgeon, incision type as well as distance between surface of removed breast and glandular tissue.
  Presence of RBT will also be assessed with regard to the distribution within the points A-O and the percentage of RBT-positive biopsies of the entity of all biopsies.

SECONDARY OUTCOMES:
Distance between surface of the removed breast and glandular tissue | 20 months
  Five additional incisions will be taken and marked on the mastectomy specimens (A2-E2), positioned in radial direction and opposite to the biopsy points A-E. The distance will be measured by the pathologist in mm.
  Outcome measurements will be the distribution of distances within the points A2-E2 (Friedman-Test), the correlation between distance points A2-E2 and corresponding biopsy points A to E as well as the correlation of the distance with RBT and with patient- and therapy-related factors (linear regression).
Detection of residual disease | 20 months
  Each biopsy specimen will be histopathologically assessed for the presence of residual disease:
  In case of SSM 10 biopsy specimens (points A-K) and in case of NSM 14 biopsy specimens (points A-O).
  The measurement of this outcome will be carried out in a descriptive way of the percentage of biopsies with residual disease, because a low number of residual disease-positive biopsies will be expected.
Correlation of patient- and therapy-related factors with residual breast tissue (RBT) and with distance between surface of removed breast and glandular tissue | 20 months
  Comparisons of patient- and therapy-related variables between SSM and NSM will be done with χ2 - and Student's t-tests for equal or unequal variances, wherever applicable. Forward-and backward logistic regression will be used to assess the influence of putative risk factors on RBT (binary dependent variable; 0: no RBT; 1: at least one probe with positive breast tissue detection). Variables will be included at P < 0.05 and excluded at P > 0.1. For all tests, statistical significance will be assumed at P ≤ 0.05.

CONTACTS AND LOCATIONS:
Locations (1):
- Brust-Zentrum AG, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papassotiropoulos B, Guth U, Chiesa F, Rageth C, Amann E, Baege A, Elfgen C, Varga Z, Moskovszky L, Endhardt K, Masser R, Tinguely M, Farhadi J, Lardi A, Dammann F, Diebold J, Li Q, Dubsky P, Tausch C. Prospective Evaluation of Residual Breast Tissue After Skin- or Nipple-Sparing Mastectomy: Results of the SKINI-Trial. Ann Surg Oncol. 2019 May;26(5):1254-1262. doi: 10.1245/s10434-019-07259-1. Epub 2019 Mar 4. PMID 30830538